CLINICAL TRIAL: NCT02153164
Title: Effect of the Steep Trendelenburg Position on Respiratory Gas Heat Content
Status: Completed | Type: Observational
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Other Study IDs: 589602
Record Dates: First submitted 2014-05-29; First posted 2014-06-02 (Estimated); Last update posted 2017-08-14 (Actual); Status verified 2017-08

CONDITIONS: Effect of Patient Position on Airway Heat Content
Keywords: Enthalpy; Trendelenberg position; Mechanical ventilation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a single site, prospective, non-blinded, non-randomized, non-interventional study designed to evaluate the effect of changes in patient position on the measurement of respiratory heat loss (enthalpy). This study would be carried out on patients whose operation requires the use of the steep Trendelenburg position independent of this study.

ELIGIBILITY:
Inclusion Criteria:

* age greater than 18 years
* scheduled for an elective surgical procedure requiring general anesthesia, positive pressure ventilation using an endotracheal tube and the steep Trendelenburg position

Exclusion Criteria:

* Adults unable to give primary consent
* age less than 18 years
* pregnancy
* prisoners
* infusion of inotropic drugs
* positive end expiratory pressure (PEEP) requirements >8 cm H2O Women, minorities or non-English speaking subjects will not be excluded.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Elective surgery requiring steep Trendelenberg position.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2015-07 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Respired gas heat content | 6 months
  (6 months for protocol and 2 hours per patient)

CONTACTS AND LOCATIONS:
Overall Officials: Neal W. Fleming, M.D., Ph.D., Principal Investigator — University of California Davis, Department of Anesthesiology and Pain Medicine